CLINICAL TRIAL: NCT01259180
Title: Efficacy of Acupuncture on Chronic Pelvic Pain in Women With Endometriosis or Adenomyosis : A Preliminary Study
Brief Title: Efficacy of Acupuncture on Chronic Pelvic Pain in Women With Endometriosis or Adenomyosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: East West Neo Medical Center (Other)
Responsible Party: Dae-Hyun Kim, East-West Neo Medical center clinical medicine institute
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KUIMS-pp-10
Record Dates: First submitted 2010-12-13; First posted 2010-12-14 (Estimated); Last update posted 2010-12-14 (Estimated); Status verified 2010-10

CONDITIONS: Endometriosis; Adenomyosis; Pelvic Pain
Keywords: acupuncture
MeSH Terms: conditions — Endometriosis; Adenomyosis; Pelvic Pain | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Acupuncture group (Experimental): twice a week, 6 weeks real acupuncture treatment, 12 sessions
  Interventions: Procedure: acupuncture treatment
- Sham acupuncture group (Sham Comparator): twice a week, 6 weeks real acupuncture treatment, 12 sessions
  Interventions: Procedure: Sham acupunture
- Control group (No Intervention): observation.

INTERVENTIONS:
Procedure: acupuncture treatment — twice a week, 6 weeks, 12sessions penetrating skin with stailess steel acupuncture device(diameter: 0.25-0.3mm,legth: 30-70mm) points: BL 23,BL31,BL32, BL40, BL53, GB30, SP 6 bilaterally plus Ashi. with
  Arms: Acupuncture group
Procedure: Sham acupunture — twice a week, 6 weeks, 12 sessions not penetrating skin with dull acupuncture device(Park Sham device :Acuprime Co. Ltd, UK) point: 1~2inches away from real acupuncture point
  Arms: Sham acupuncture group

SUMMARY:
The purpose of ths study is to determine the efficacy of acupuncture on chronic pelvic pain in women with endometriosis or adenomyosis.

DETAILED DESCRIPTION:
Chronic pelvic pain(CPP) is a common disease among women, and its prevalence ranges from 4 to 25 percent. There are various conditions associated with CPP, including gynecologic, urologic and gastointestinal problems. Endometriosis is the most common diagnosis made at the time of gynecological laparoscopy performed to evaluate CPP. Treatments of CPP with endometriosis include medical(analgesics, oral contraceptive pills, gonadotropin releasing hormone(GnRH) agonist, etc.), surgical and combined treatment. Progestins, danazol, estrogen-progestin pills, or GnRH agonists are commonly used as a concurrent treatment along with surgery. However, a systematic review on the comparison of postsurgical hormonal suppression to surgery alone concluded that, while postoperative medical therapy decreased recurrence rates, there was no significant benefit on the outcomes of pain and pregnancy rates. Therefore there is a need for postoperaive medical therapy for pain relief. In this study, the investigators propose a randomized, sham-controlled trial to investigate the efficacy of acupuncture as a pain control for the patients dignosed endometriosis during laparoscopic surgery due to CPP, and have been on 6 month-scheduled GnRH agonist treatment as a postoperative treatment.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed pathologically of Endometriosis or Adenomyosis among those who had undergone laparoscopic surgery due to pelvic pain
* Patients who have been on GnRH agonist treatment for 6 months after being diagnosed Endometriosis or Adenomyosis
* Patients who agreed a written consent by their own will
* Patients' compliance and geographical adjacency appropriate for proper follow up survey
* continuous pelvic pain over VAS 5 during past 1 week on screening visit(after 6 weeks of surgery) (0='no pain', '10=most severe')

Exclusion Criteria:

* Those who had taken hormones or drugs that can affect diagnosis of endometriosis or adenomyosis for past 1 year
* Patients found to have malignant tumor of uterus and adenexa, PID or pregnancy during surgery
* Allergies to metal or contraindications for acupuncture treatment (ex: coagulopathy, epilepsy)
* Unable to participate in clinical trial by doctor's judgment
* irritable bowel syndrome

Ages: 16 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-09 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
Chages in Visual Analogue Scale of subjective Pelvic Pain | 7wks

SECONDARY OUTCOMES:
Health-related Quality of Life | 7wks
  1.36-item Short-Form Health Survey Version 2.0 2.Beck's Depression Index 3.Social Readjustment Rating Scale 4. Heart Rate Variability 5. Digital Infrared Thermographic Image 6. Assessment of Voice

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Moo Lee, OMD, Study Director — East West Neo Medical Center
Locations (1):
- East-West Neo Medical Center, Seoul, Seoul, South Korea